CLINICAL TRIAL: NCT00757796
Title: Obstructive Sleep Apnea Syndrome and Attention Executive Function Disturbances
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Itzhak Shpirer, The Sleep Laboratory, Assaf Harofeh Medical Center, Zerifin, Israel
Other Study IDs: 143/06
Record Dates: First submitted 2008-09-21; First posted 2008-09-23 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Studies demonstrate that sleep disturbances are associated with cognitive dysfunction and attention deficit. However the correlation between the severity of obstructive sleep apnea and the degree of cognitive dysfunction was not demonstrated. Our hypothesis is that patients suffering from a more severe sleep apnea will demonstrate a greater degree of cognitive dysfunction.

DETAILED DESCRIPTION:
Studies demonstrate that sleep disturbances are associated with cognitive dysfunction and attention deficit. However the correlation between the severity of sleep disturbances and the degree of cognitive dysfunction was not demonstrated.We intend to study 80 patients with various degrees of obstructive sleep apnea. All patients will undergo executive cognitive tests as well as tests to assess for levels of depression, anxiety and attention.

ELIGIBILITY:
Inclusion Criteria:

1. Apnea hypopnea index>5
2. Age 20 - 70 years

Exclusion Criteria:

1. Pregnant women
2. Known chronic cardiovascular or pulmonary disease
3. Patients s/p CVA or brain damage
4. Known depression or other psychiatric disorder
5. Patients with severe cognitive dysfunction (MMSE<25)
6. Patients receiving stimulants, antipsychotic or anti-depression medications

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 20 - 70 years with obstructive sleep apnea.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-10